CLINICAL TRIAL: NCT06825104
Title: Long-Term Evaluation of TAILORED Vs Anatomical Ablation Strategy for Persistent Atrial Fibrillation
Acronym: TAILORED-LT
Status: Recruiting | Type: Observational
Sponsor: Volta Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIPL-01-006
Record Dates: First submitted 2025-01-31; First posted 2025-02-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
Keywords: Artificial Intelligence; VX1; Volta AF-Xplorer; Medical Device; Cardiac Dispersion; Volta Medical; Software
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Experimental: Tailored: Patients from the "Tailored" group in the initial study TAILORED-AF. Patients in this group underwent "Tailored" AF ablation, i.e. the analysis and targeting of pathological areas using Volta Medical's artificial intelligence software (Volta AF-Xplorer, formerly VX1), in addition to electrical isolation of the pulmonary veins (PVI).
  Interventions: Device: Volta AF-Xplorer; Procedure: Dispersion ablation + PVI
- Active Comparator: Anatomical: Patients from the "Anatomical" group in the initial study TAILORED-AF. Patients in this group underwent PVI only.
  Interventions: Procedure: PVI

INTERVENTIONS:
Device: Volta AF-Xplorer — Dispersion ablation strategy guided by Volta Medical AI-software targeting areas of spatiotemporal dispersed electrograms
  Groups: Experimental: Tailored
Procedure: Dispersion ablation + PVI — TAILORED-AF index procedure: Dispersion ablation + PVI
  Groups: Experimental: Tailored
Procedure: PVI — TAILORED-AF index procedure: PVI only
  Groups: Active Comparator: Anatomical

SUMMARY:
The TAILORED-LT study is conducted as an extension follow-up until 5 years of the initial TAILORED-AF study (NCT04702451), in order to demonstrate the long-term superiority in terms of freedom of atrial fibrillation (AF) of a tailored ablation strategy targeting areas of spatio-temporal dispersed electrograms in combination with pulmonary veins isolation (PVI) over an anatomical ablation strategy targeting PVI alone for the initial ablation procedure of persistent AF.

DETAILED DESCRIPTION:
The TAILORED-AF study demonstrated at one year's follow-up that a tailored ablation strategy guided by Volta Medical AI-software targeting areas of spatio-temporal dispersed electrograms in combination with pulmonary vein isolation (PVI) ablation is more effective to an anatomical ablation strategy targeting PVI alone (current standard of care) for the treatment of persistent atrial fibrillation (AF).

VX1 legacy device renamed Volta AF-Xplorer was used in the TAILORED-AF study in the treatment arm.

No additional treatments are specifically required in the scope of this ancillary TAILORED-LT study which aims to follow the patients previously treated in the initial TAILORED-AF study over the long-term. However, in the event of repeat procedures during the TAILORED-LT study, the choice of the ablation technique will be left to the investigator's discretion, regardless of the patient's randomization arm in the TAILORED-AF study.

The annual follow-up will be performed as in routine clinical practice post AF ablation procedures: visits at 24 months, 36 months, 48 months and 60 months post TAILORED-AF Study index procedure. It is possible that some of these annual visits cannot be completed prospectively due to time already having elapsed between the end of the subject participation in the TAILORED-AF study and the date of enrollment in the extension TAILORED-LT study. In this case, available data (among those expected by the study protocol) will be collected retrospectively.

The additional procedures related to this clinical investigation are limited to annual 24-hour Holters and to the administration of Quality Of Life questionnaires (SF-36 and AFEQT) to the patients during follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patient who participated in the Tailored AF study
* Patient not withdrawn during the 12-month follow-up period post-index procedure in the Tailored AF study
* Patient able and willing to provide written informed consent to participate in this extension Tailored-LT study

Exclusion Criteria:

* Person deprived of liberty or under guardianship
* Person unable to undergo a medical monitoring for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients previously enrolled in TAILORED-AF study, treated for their persistent AF by an index ablation procedure and not withdrawn during the 12-month follow-up period post-index procedure.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Long-term freedom from documented atrial fibrillation (AF) after one ablation procedure | 60 months
  Long-term freedom from documented AF episodes > 30 seconds, with or without antiarrhythmic drugs (AADs), after a single index ablation procedure.

SECONDARY OUTCOMES:
Long-term freedom from documented AF/AT after one or two ablation procedures | 60 months
  Long-term freedom from documented AF and Atrial Tachycardia (AT) episodes > 30 seconds, after one or two procedures, with or without AADs
Long-term freedom from documented AF/AT after one ablation procedure | 60 months
  Long-term freedom from documented AF/AT episodes > 30 seconds, after one procedure, with or without AADs
Heath Economics - Average Number of Ablation Procedures per patient | 60 months
  To determine how the number of repeat ablation procedures in addition to the index procedure impacts health care costs.
Heath Economics - Average Number of Hospitalizations per patient | 60 months
  To determine how the number of hospitalizations post-ablation index procedure impacts health care costs.
Heath Economics - Average Number of Cardioversions per patient | 60 months
  To determine how the number of cardioversions post-ablation index procedure affects health care costs.
Heath Economics - Quality of Life Progression (AFEQT Score) | 60 months
  To determine how the quality of life progression after the ablation index procedure (measured with the Atrial Fibrillation Effect on Quality of Life Questionnaire AFEQT) impacts health care costs.
  AFEQT score ranges from 0 to 100, with higher scores indicating better quality of life.
Heath Economics - Quality of Life Progression (SF-36 Score) | 60 months
  To determine how the Quality of life progression after the ablation index procedure (measured with the 36-Item Short Form Health Survey SF-36) impacts health care costs.
  The SF-36 consists of eight domains measuring physical and mental health, with scores ranging from 0 to 100 (higher scores indicate better quality of life).
Heath Economics - Proportion of Patients Under AAD | 60 months
  To determine how the proportion of patients under antiarrhythmic drugs (AAD) impacts health care costs.
Incidence of complications (safety composite endpoint) | 60 months
  Incidence of complications: death, cerebrovascular events, or serious treatment-related adverse event at long-term.
  NOTE: In addition, each component of the composite endpoint will be individually assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel DEISENHOFER, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (13):
- France (11):
  - CHU Lyon, Hôpital Louis Pradel, Bron
  - Pôle Santé République, Clermont-Ferrand
  - Hôpital Saint Philibert, Lomme
  - Hôpital Saint-Joseph Marseille, Marseille
  - Hôpital Privé Jacques Cartier, Massy
  - Hôpital Privé du Confluent, Nantes
  - Polyclinique Saint George, Nice
  - Centre Cardiologique du Nord, Saint-Denis
  - Clinique Rhéna, Strasbourg
  - Clinique Pasteur, Toulouse
  - CHRU Nancy, Institut Lorrain du coeur et des vaisseaux, Vandœuvre-lès-Nancy
- Germany (2):
  - Klinikum Coburg, Coburg
  - German Heart Center, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deisenhofer I, Albenque JP, Busch S, Gitenay E, Mountantonakis SE, Roux A, Horvilleur J, Bakouboula B, Oza S, Abbey S, Theodore G, Lepillier A, Guyomar Y, Bessiere F, Jan Smit J, Mohr Durdez T, Milpied P, Appetiti A, Guerrero D, De Potter T, De Chillou C, Goldbarg S, Verma A, Hummel JD; TAILORED-AF Investigators. Artificial intelligence for individualized treatment of persistent atrial fibrillation: a randomized controlled trial. Nat Med. 2025 Apr;31(4):1286-1293. doi: 10.1038/s41591-025-03517-w. Epub 2025 Feb 14. PMID 39953289
- [Background] Seitz J, Bars C, Theodore G, Beurtheret S, Lellouche N, Bremondy M, Ferracci A, Faure J, Penaranda G, Yamazaki M, Avula UM, Curel L, Siame S, Berenfeld O, Pisapia A, Kalifa J. AF Ablation Guided by Spatiotemporal Electrogram Dispersion Without Pulmonary Vein Isolation: A Wholly Patient-Tailored Approach. J Am Coll Cardiol. 2017 Jan 24;69(3):303-321. doi: 10.1016/j.jacc.2016.10.065. PMID 28104073
- [Background] Seitz J, Durdez TM, Albenque JP, Pisapia A, Gitenay E, Durand C, Monteau J, Moubarak G, Theodore G, Lepillier A, Zhao A, Bremondy M, Maluski A, Cauchemez B, Combes S, Guyomar Y, Heuls S, Thomas O, Penaranda G, Siame S, Appetiti A, Milpied P, Bars C, Kalifa J. Artificial intelligence software standardizes electrogram-based ablation outcome for persistent atrial fibrillation. J Cardiovasc Electrophysiol. 2022 Nov;33(11):2250-2260. doi: 10.1111/jce.15657. Epub 2022 Sep 18. PMID 35989543